CLINICAL TRIAL: NCT04253444
Title: A Randomized Single Blinded Parallel Study to Investigate the Physiological Modulation of the Autonomic Nervous System on Symptoms in Patients With Reflux Hypersensitivity
Brief Title: The Effect of Autonomic Modulation on Symptoms in Patients With Reflux Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 278533
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-10

CONDITIONS: Gastro Esophageal Reflux
Keywords: slow deep breathing; vagal nerve stimulation; reflux hypersensitivity
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: A randomised, sham-controlled, single-blinded, parallel study
Who Masked: Participant
Masking Description: Participants and outcomes assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- slow deep breathing (Active Comparator): Patients are instructed to do deep breathing at full inspiratory capacity for 4 seconds followed by forced expiration in 6 seconds (forced vital capacity) for 10 minutes.
  Interventions: Behavioral: slow deep breathing
- sham breathing (Sham Comparator): Patients are instructed to count 10 breaths and tick a box every time they count ten breaths. The counting distracts the patient reducing the effect of focussing of breathing on their autonomic nervous system.
  Interventions: Behavioral: sham breathing

INTERVENTIONS:
Behavioral: slow deep breathing — Participants in this arm will be asked to do slow deep breathing (4 seconds inhalation and 6 seconds exhalation) for 10 minutes twice a day during the study period.
  Arms: slow deep breathing
Behavioral: sham breathing — Participants in this arm will be asked to do sham breathing for 10 minutes twice a day during the study period.
  Arms: sham breathing

SUMMARY:
Reflux hypersensitivity is the disease that causes chest pain, heartburn and regurgitation and can impair patients' quality of life. Pain modulators are often used for the treatment of reflux hypersensitivity, but the effect is not enough and more effective therapy is needed.

Slow deep breathing is the validated method to modulate the autonomic nervous system. In our previous study, slow deep breathing could increase the threshold of oesophageal pain in healthy volunteers. Therefore, slow deep breathing has the potential to be an effective treatment for reflux hypersensitivity and further study is warranted in the patient group.

The aims of this study are (1) to evaluate the feasibility of slow deep breathing and (2) to investigate the effect of autonomic nerve modulation by slow deep breathing on symptoms in patients with reflux hypersensitivity.

DETAILED DESCRIPTION:
This is a randomized single-blinded parallel study and the investigators aim to recruit 40 participants.

Patients will be enrolled for a period of 4 weeks and don't have to attend our institution. A video chat on day 1 will consist of confirming eligibility, after which the patient will be randomised to follow either the slow deep breathing protocol or the sham breathing protocol in a single blinded fashion. That is, the patient will be unaware of which the active breathing exercise is. Once randomised during a video chat, they will undergo baseline heart rate variability (HRV) measurements using a smartphone app, answer the questionnaires on Research Electronic Data Capture (REDCap), and then practice the relevant breathing exercise with an instruction video. The patient will then be trained to self-administer the breathing exercise during a video chat, which will be used twice a day for 10 minutes over the next 4 weeks with a standardized instruction video.

This study finishes when participants answer the online questionnaire and record HRV on day 29.

The investigators will set up this questionnaire on our electronic data capture system (Research Electronic Data Capture: REDCap). Participants will answer questionnaires using this online system on day 1, day 8, day15, day 22, and day 29 (end of the study).

Therefore, participants will also be trained on how to use REDCap and answer questionnaires under supervision on day 1 during a video chat. Questionnaires on day 8, 15, 22, and 29 will be answered at home. The investigators will send a reminder message to participants using a REDCap system the day before they answer the questionnaire.

Participants will be asked to record their HRV using a smartphone app on day 1, 8, 15, 22, and 29.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 18 years.
* Women in the follicular phase of the menstrual cycle (visits will be arranged so that in menstruating women, the study will be started in the follicular phase of the menstrual cycle to standardise for possible confounding effects of the menstrual cycle on symptom perception).
* Able to give informed consent
* Able to speak and understand English without the need for an interpreter
* No evidence of erosive esophagitis by OGD
* Presence of chest pain, heartburn, and/or regurgitation ≥ 3 days/week
* Normal acid exposure on MII-pH
* Positive symptom reflux association on MII-pH (symptom index ≥ 50% and symptom association probability ≥ 95%)
* OGD is performed within 2 years before the enrolment
* MII-pH study is performed within 2 year before the enrolment

Exclusion Criteria:

* Current or previous GI or medical illnesses that may affect ANS / GI function
* Current or previous significant CNS illness
* Current medications affecting the CNS, GI or ANS systems
* Pregnancy and lactation
* Cardiac dysrhythmias
* Those who do not have access to the internet-based questionnaire

  * The use of acid suppression therapies (e.g. proton pump inhibitor or H2 blocker) or pain modulators (e.g. low-dose Tricyclic Antidepressants, TCAs or Selective Serotonin Reuptake Inhibitors, SSRI) does not change the decision of participation as long as above-mentioned symptoms remain.

Patients are asked to refrain from smoking for 12 hours and drinking alcohol as well as using recreational drugs for 48 hours prior to study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The feasibility of 10 minutes twice a day for 4 weeks of slow deep breathing | 4 weeks
  Compliance and acceptability are evaluated by the Global or general acceptability of treatment questionnaire. This is recorded as 'very good', 'good', 'fair', or 'poor'.

SECONDARY OUTCOMES:
The effect of slow deep breathing on anxiety | 4 weeks
  State and Trait Anxiety Inventory state (Maximun and minimum values are 80 and 20, respectively. The higher value indicates more nervous status.) and State and Trait Anxiety Inventory trait (Maximun and minimum values are 80 and 20, respectively. The higher value indicates more nervous trait) are used.
The effect of slow deep breathing on personality states. | 4 weeks
  Big five inventory questionnaire (44 items) is used. This is a self-report inventory designed to measure the personality type.
The effect of slow deep breathing on depression. | 4 weeks
  Hospital Anxiety and Depression Scale is used. The maximun and minimum values are 21 and 0, respectively (0-7 = Normal, 8-10 = Borderline,11-21 = Abnormal).
Changes in vagal nerve activity before and after slow deep breathing protocol | 4 weeks
  Cardiac vagal tone, which is an indicator of vagal nerve activity and caluculated from R-R interval of electrocardiogram, is used for the evaluation.
Changes in symptoms before and after slow deep breathing | 4 weeks
  Reflux symptom questionnaire, 7 day recall is used for the evaluation. This can categorize the symptom into 'did not have', 'very mild', 'mild', 'moderate', 'moderately severe', or 'severe'.

CONTACTS AND LOCATIONS:
Overall Officials: Qasim Aziz, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No